CLINICAL TRIAL: NCT02014922
Title: A Study to Determine the Relief of Dry Eye Symptoms With the Use of TheraTears® Products
Brief Title: A Study to Determine the Relief of Dry Eye Symptoms With the Use of TheraTears® Products (DUNLIN)
Acronym: DUNLIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Advanced Vision Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P/439/13/AVR
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants randomized to the control group will be allowed to continue using their habitual artificial tears, and / or additional habitual concurrent dry eye treatments.
- Treatment (Experimental): Participants in the study treatment group will receive all four products:
  * TheraTears® Lubricant Eye Drop (15mL) - Dosage: Ophthalmic, 1 or 2 drops, prn
  * TheraTears® preservative-free single-use containers (32-pack, 0.6mL each) - Dosage: Ophthalmic, 1 or 2 drops, prn
  * TheraTears® Nutrition (90 pack) - Dosage: Oral, 3 capsules QD
  * TheraTears® TheraLid® Eyelid Cleanser (48mL) - Dosage: Ophthalmic, 1 or 2 application OU, QD
  Interventions: Drug: TheraTears® Lubricant Eye Drop; Drug: TheraTears® preservative-free single-use containers; Dietary Supplement: TheraTears® Nutrition; Other: TheraTears® TheraLid® Eyelid Cleanser

INTERVENTIONS:
Drug: TheraTears® Lubricant Eye Drop
  Arms: Treatment
Drug: TheraTears® preservative-free single-use containers
  Arms: Treatment
Dietary Supplement: TheraTears® Nutrition
  Arms: Treatment
Other: TheraTears® TheraLid® Eyelid Cleanser
  Arms: Treatment

SUMMARY:
Dry eye is a very common condition that most often affects women and the elderly, and can be caused when the eyes do not produce enough tears, or when the tears evaporate too quickly. Although there isn't a simple cure for dry eye, there are numerous products on the market that attempt to help relieve some of the discomfort caused by this condition. Some of these products include artificial tears, omega-3 supplements, and/or anti-inflammatory medications. The purpose of this study is to evaluate the performance of a combination of TheraTears® products, and to compare them with the product(s) you have been using.

ELIGIBILITY:
Inclusion Criteria:

1. Is between 18 and 65 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Exhibits symptoms of dry eye for at least 3 months;
5. Has an OSDI score of ≥ 23;
6. Is currently on a non-omega 3 dry eye treatment regimen that, at the minimum consists of instilling artificial tears at least once a day for the past 3 months;
7. Has an average non-invasive tear breakup time ≤ 5.00 seconds in at least one eye.

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection and/or allergies;

   * For the purposes of study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are typical findings and are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Is pregnant, lactating or planning a pregnancy at the time of enrollment, as determined verbally;
7. Is aphakic;
8. Has undergone refractive error surgery;
9. Has taken part in another (pharmaceutical) research study within the last 30 days;
10. Has worn contact lenses within the past 5 years;
11. Is currently using or have used omega 3 supplements in the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change over time of OSDI score | At screening, 2 weeks, 1 month and 3 months
  Ocular Surface Disease Index (OSDI) questionnaire score
Change over time of Visual analogue scores | At screening, 2 weeks, 1 month and 3 months
Change over time of Tear osmolarity | At screening, 1 month and 3 months
Change over time of Tear film breakup time | At screening, 1 month and 3 months
Change over time of Corneal staining | At screening, 1 month and 3 months

SECONDARY OUTCOMES:
Change over time of Lid wiper epitheliopathy | At screening, 1 month and 3 months
Change over time of Meibomian gland expressibility | At screening, 1 month and 3 months
Change over time of Meibum quality | At screening, 1 month and 3 months
Change over time of Tear film lipid layer thickness | At screening, 1 month and 3 months
Change over time of Tear meniscus height | At screening, 1 month and 3 months
Change over time of Schirmer's I scores | At screening, 1 month and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Contact Lens Research, University of Waterloo School of Optometry & Vision Science, Waterloo, Ontario, Canada